CLINICAL TRIAL: NCT04135456
Title: Study on the Optimal Dosage of Mannitol in Aneurysmal Subarachnoid Hemorrhage Craniotomy
Brief Title: The Optimal Dose of Mannitol for Intraoperative Brain Relaxation During the Operation of Aneurysmal Subarachnoid Hemorrhage
Acronym: ODAS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Wang Shuo, Director of Department of Cerebrovascular Neurosurgery, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY 2019-09
Record Dates: First submitted 2019-09-11; First posted 2019-10-22 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Mannitol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose group (Experimental): 0.5g/kg of 20% mannitol administered at skin incision.
  Interventions: Drug: Mannitol
- Medium dose group (Experimental): 1.0g/kg of 20% mannitol administered at skin incision.
  Interventions: Drug: Mannitol
- High dose group (Experimental): 1.5g/kg of 20% mannitol administered at skin incision.
  Interventions: Drug: Mannitol

INTERVENTIONS:
Drug: Mannitol — When the neurosurgeon starts the skin incision, 20% mannitol administered through the venous catheter with fulldrip in 5-10 minutes. Neurosurgeons evaluate the degree of brain relaxation after dura opening in 4 point scale (1=bulging brain, 2=firm brain, 3=satisfactorily relaxed, 4=perfectly relaxed).

SUMMARY:
Aneurysmal subarachnoid hemorrhage (aSAH) tended to lead to a sudden increase in intracerebral pressure (ICP), which can cause decreased cerebral perfusion and transient global cerebral ischemia. Early clipping and coiling of aneurysms and surgical evacuation of intracerebral hematoma were recommended for aSAH patients. However, the high ICP made it difficult to separate the subarachnoid space during the operation. Effective reduction of ICP was the key to the succession of the operation. But there is a lack of consensus on the management of raised ICP in aSAH. Mannitol is widely used to reduce ICP in patients with cerebral edema. The potential mechanism including decreasing the viscosity of the blood improving regional cerebral microvascular flow and oxygenation and increasing intravascular volume due to increased plasma osmolality. The magnitude of the pressure reduction was correlated with the intact intracranial automatic adjustment function. However, the hypochloremic metabolic alkalosis, hypernatremia, hypokalemia and renal failure associated with mannitol overdose must be considered and the effective dose and the duration of its administration were still unknown. The aims of this study were to determine the most appropriate mannitol dose to provide adequate brain relaxation in aSAH patients with the fewest adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute subarachnoid hemorrhage
* Patients who underwent frontal-temporal craniotomy pterional approach aneurysm clipping surgery under general anesthesia.
* Patients operated by the same surgeon (Dr. Chen Xiaolin).

Exclusion Criteria:

* Patients who do not agree to the surgery.
* Patients who have congestive heart failure and kidney insufficiency.
* Patients who have pre-operative electrolyte imbalance.
* Patients who did not take the frontotemporal pterygoid approach.
* Patients with contraindications to mannitol due to low blood pressure.
* Patients who have had more than 3 days from bleeding to surgery.
* Patients with intracranial hematoma.
* Patients with Hunt-Hess grades 4-5.
* Patients who received intravenous mannitol within 6 hours before surgery.
* Patients who underwent ventricle puncture and drainage surgery before surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2024-01-14 (Estimated)

PRIMARY OUTCOMES:
Brain relaxation score | Intraoperative
  The degree of brain relaxation after administration was assessed as four grades.
  denoting bulging or the condition that additional methods for brain relaxation are immediately and always required in order to continue the surgical procedure because of brain swelling; firm or the condition that additional methods for brain relaxation are occasionally required to continue the surgical procedure; adequate; perfectly relaxed. All patients received conventional frontotemporal pterional approach, and the time from skin incision to dural opening was constant for 30 minutes. At the time of dural opening, the degree of cerebral relaxation was evaluated, and the satisfactory cerebral relaxation was defined as 3 or 4 points.

SECONDARY OUTCOMES:
electrolyte change (potassium) | before the infusion of mannitol and 30 minutes after the administration of the study drug.
  Check the serum laboratory result of potassium (normal range: 3.4-4.5 mmol/L)
electrolyte change (sodium) | before the infusion of mannitol and 30 minutes after the administration of the study drug.
  Check the serum laboratory result of sodium (normal range: 136-146 mmol/L)
electrolyte change (chlorine) | before the infusion of mannitol and 30 minutes after the administration of the study drug.
  Check the serum laboratory result of chlorine (normal range: 98-106 mmol/L)
electrolyte change (calcium) | before the infusion of mannitol and 30 minutes after the administration of the study drug.
  Check the serum laboratory result of calcium (normal range: 1.15-1.29 mmol/L)
Subdural hematoma | CT scan 6 hours after surgery
  Excessive decrease in intracranial pressure may lead to intraoperative or postoperative subdural hematoma formation
modified Rankin Score 3 months after surgery | 3 months after surgery
  To evaluate the potential benefits of effective dural lysis and brain relaxation on patient outcomes. The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms. 1 - No significant disability. Able to carry out all usual activities, despite some symptoms. 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities. 3 - Moderate disability. Requires some help, but able to walk unassisted. 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Dead.

OTHER OUTCOMES:
operation duration | intraoperative
  Poor intracranial pressure reduction may result in prolonged duration of surgery, and evaluation of the duration of surgery is helpful in the selection of the optimal dose.Poor intracranial pressure reduction may result in prolonged duration of surgery, and evaluation of the duration of surgery is helpful in the selection of the optimal dose.

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Wang, MD, Principal Investigator — Beijing Tiantan Hospital; Xiaolin Chen, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Capital Medical University Affiliated Beijing Tiantan Hospital, Beijing, Beijing Municipality, China